CLINICAL TRIAL: NCT01433718
Title: The Effectiveness of Neuromuscular Training on Modifiable Anterior Cruciate Ligament Injury Risk Factors
Brief Title: Decreasing Knee Injury Risk Factors With Neuromuscular Training
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Athletic Trainers' Association Research & Education Foundation (NATA Foundation) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ohio_U11F024; 1104MGP005 (Other Grant/Funding Number: National Athletic Trainers' Association Research & Education Foundation)
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: ACL; Anterior Cruciate Ligament Injury
Keywords: Effectivness; Neuromuscular Training; Resistance Training; Modification; Anterior Cruciate Ligament Risk Factors; Drop-Jump; Knee Separation; Resistance training program
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACL prevention training (Experimental)
  Interventions: Procedure: Neuromuscular and Resistance Training

INTERVENTIONS:
Procedure: Neuromuscular and Resistance Training — 1 hour/session, 3 sessions/week, 6 weeks

SUMMARY:
Anterior cruciate ligament (ACL) tears are disabling injuries that place a significant burden on the athlete. Roughly 80% of these injuries are linked to a noncontact mechanism, with more than 70% of them occurring while landing from a jump. Female athletes are at higher risk of sustaining a noncontact ACL injury due to the higher number of risk factors that they possess compared to their male counterparts. Due to this statistic, ACL prevention programs have been developed over the past 15 years in attempt to reduce this risk among the female athletic population. These programs have been shown to reduce the rate of noncontact ACL injuries in females by correcting the risk factors associated with them. However, it remains unclear as to whether these positive results are solely due to the program or a higher exercise workload in its participants. The purpose of this study is to evaluate the effectiveness that an ACL prevention program has on modifying at-risk landing mechanics (associated with noncontact ACL injury) compared to a resistance training program of equal workload.

DETAILED DESCRIPTION:
Injury Background Anterior cruciate ligament (ACL) tears are disabling injuries that place a significant burden on the athlete. The average cost for ACL reconstruction is estimated to be approximately $17,000 per patient and full recovery commonly takes around 6 months to achieve. It has been estimated that 1 in every 3000 people in the United States suffer an ACL rupture each year. Roughly 80% of these injuries are linked to a noncontact mechanism, with more than 70% of them occurring while landing from a jump.

Injury Mechanism Upon landing, the lower body falls into what is referred to as the "position-of-no-return" (PNR). The landing kinematics involved with the PNR places a high amount of stress on the ACL and can ultimately lead to a complete rupture.

Injury Imbalance Female athletes who participate in sports that involve jumping and cutting activities suffer 4-to-6 times more ACL injuries than males who participate in the same sports. This is attributed to the higher number of risk factors that females possess during and after puberty. In particular, upon maturation, males exhibit a neuromuscular spurt, with increases in power, strength, and coordination, whereas females do not. Other risk factors that females demonstrate are quadriceps dominance and ligament dominance. Both of these dominances are linked to the landing kinematics of the knee when placed in the PNR.

Quadriceps dominance is characterized by the extended knee posture that is displayed in the PNR when landing from a jump. When landing on an extended knee, the tibia is translated anteriorly to the femur, causing the ACL to become taunt. In order to prevent the ACL from rupturing, the hamstrings must activate to flex the knee and translate the tibia posteriorly. In response to anterior tibial translation, females are found to utilize a different muscle recruitment pattern than males by contracting their quadriceps before their hamstrings, whereas males follow the opposite pattern. By contracting the quadriceps first, the hamstrings are overpowered, which allows for further anterior tibial translation to occur during landing.

Ligament dominance is evidenced by the increased knee valgus that displayed in the PNR when landing and cutting. During these maneuvers, females rely on their knee ligaments rather than lower extremity musculature to absorb ground reaction forces. This tendency places a high amount of stress on the ACL, which in turn, increases the probability of it rupturing.

Injury Prevention Due to the high rate of noncontact ACL injuries seen in female athletes, neuromuscular training (NMT) programs have been developed in an attempt to prevent or reduce the risk of injury. These programs are administered as either an off-season regimen or in-season warm-up routine, and they incorporate a combination of plyometric, proprioceptive, and strength training exercises, with particular focus being placed on correct technique. By modifying neuromuscular risk factors, NMT programs have been able to significantly reduce the rate of noncontact ACL injury.

Specific Aim 1:

To evaluate the effectiveness that an ACL prevention program has on modifying at-risk landing mechanics (associated with noncontact ACL injury) compared to a resistance training program of equal workload.

Specific Aim 2:

To evaluate the effectiveness that an ACL prevention program has on improving max vertical jump height compared to a resistance training program of equal workload.

ELIGIBILITY:
Inclusion Criteria:

* Female college underclassman (ages 18-20)
* Body Mass Index (BM) between 18.5 - 25 (normal range)
* Blood pressure below 140/90 (below hypertension)
* History of participation in high school athletics
* Signed Informed Consent form

Exclusion Criteria:

* History of ACL injury
* Current/ongoing knee condition
* History of surgical intervention within one year (not including facial)
* Current/ongoing musculoskeletal injury
* History of previous ACL prevention training
* Currently involved in intercollegiate athletics
* Currently Pregnant

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change in Knee separation during the Drop Jump Test | 1 week prior to training begins, and 1 week after training finishes.
  Participants will begin the test by standing on a box, dropping off, landing straight in front of the box, and immediately performing a maximum vertical jump. Following the completion of the three trials, the examiner chooses the trial in which the participant has the highest jump to best represent the participant's jumping ability for video analysis. The following images will be captured as still photographs: (1) pre-landing; (2) land; and (3) takeoff.

SECONDARY OUTCOMES:
Changes in Vertical Jump Test | 1 week prior to training begins, and 1 week after training finishes
  Each participant's standing reach will be recorded prior to performing the test. The participants will perform three trials, with the highest jump height being recorded. Participants will begin the test by standing directly underneath the Vertec markers and jumping vertically while reaching with their hand to swipe the highest marker possible. Arm swing will be allowed for the jump, but an approach-step will not.

CONTACTS AND LOCATIONS:
Overall Officials: Conrad M Gabler, B.S., Principal Investigator — Graduate Athletic Training Student; Brian G Ragan, Ph.D., Study Director — Athletic Training Program Assistant Professor and Research Coordinator
Locations (1):
- Ohio University, Athens, Ohio, United States